CLINICAL TRIAL: NCT03115814
Title: Deep Brain Stimulation for Treatment of Severe Alzheimer's Disease: Study Protocol of a Prospective, Self-control Phase I Trial
Brief Title: Deep Brain Stimulation for Treatment of Severe Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhiqi Mao, Principal Investigator, Chinese PLA General Hospital
Other Study IDs: ChinaPLAGH_MZQ
Record Dates: First submitted 2017-04-07; First posted 2017-04-14 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the safety of deep brain stimulation in the treatment of severe Alzheimer's disease (AD); to investigate the effectiveness of deep brain stimulation in the treatment of severe AD, i.e., effects of deep brain stimulation on cognitive function in patients with severe AD and dementia grading; to investigate the effects of deep brain stimulation on cerebral glucose metabolism in patients with severe AD.

DETAILED DESCRIPTION:
This study is a prospective, self-control, phase I trial, which will be performed in Department of Neurosurgery, Chinese PLA General Hospital (Beijing, China). Six patients with severe Alzheimer's disease will be included in this study and receive continuous bilateral deep brain stimulation of the fornix.

BACKGROUND With the prolongation of life expectancy of the world population, Alzheimer's disease (AD) has become one of the major diseases that influence the quality of life in the aging population. The latest data have shown that there are approximately 24 million AD victims and the number increases in fold every 20 years. With global population aging, there is an increasing number of population who are at the risk of AD. Epidemiological studies in China have shown that the incidence of AD increases with aging and it is about 5% in people aged over 65 years and about 20% in people aged over 85 years. AD has been reported to greatly affect patient's quality of life. However, there is currently no effective method to hinder, postpone or treat AD. Cholinesterase inhibitors (Donepezil, Galantamine and Rivastigmine) and N-methyl-D-asparate receptor antagonist Memantine are the commonly used drugs. But the curative effects are not identified. Therefore, there is an urgent need to investigate a novel treatment method of AD.

Deep brain stimulation is hopeful in the treatment of AD. There is clinical evidence that deep brain stimulation can effectively postpone, hinder and even reverse the progression of AD. The clinical data also shows that selective atrophy of cholinergic neurons of the nucleus basalis of Meynert (NBM) is one of characteristics of AD. In 1985, Turnbull et al., were the first to report the role of deep brain stimulation of the NBM in AD patients. They detected cortical glucose metabolic activity using FDG-PRT and found that the cortical glucose metabolic activity in the frontal lobe, temporal lobe, parietal lobe, and occipital lobe of the right hemisphere (not stimulated) of AD patients was decreased by 21%, 24%, 10%, and 7.5%, respectively. By contrast, cortical glucose metabolic activity in the left hemisphere was decreased by 12%, 4%, 0 and -1.5% respectively. Although there were no improvements in clinical symptoms, study findings suggest that deep brain stimulation of the NBM is safe and leads to strong pathophysiologic response. Laxton et al. performed deep brain stimulation of the hypothalamus and fornix in six patients with mild AD. At 6 and 12 months after deep brain stimulation, Mini-Mental State Examination (MMSE) and Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) evaluations showed that patient's cognitive was improved. In the same case cohort, Smith et al. investigated cerebral glucose metabolism and found that deep brain metabolism increased cerebral glucose metabolism mainly through two orthogonal networks: a frontal-temporal-parietal-striatal- thalamic network and a frontal-temporal-parietal-occipital-hippocampal network. Fontaine et al. performed deep brain stimulation in one AD patients presenting with mild cognitive disorder. Twelve months after deep brain stimulation, cerebral glucose metabolism was slightly increased in the cerebrum, in particular in bilateral middle temporal gyri; in addition, cognitive function was improved as confirmed by MMSE and ADAS-Cog evaluations.

Deep brain stimulation for treatment of AD is internationally in its infancy. Only exploratory studies involving a few cases have been reported. Similar reports are not reported in China. Global doctors eager to understand the exact effects and possible complications and risks of deep brain stimulation in the treatment of AD. AD patients are also looking forward to the effectiveness of this therapy in reducing their sufferings.

Adverse events

1. At 6 months after surgery, radiological examination of the implants will be performed to determine that the stimulation system is not impaired.
2. Deep brain stimulation parameters: frequency, amplitude and pulse width
3. After deep brain stimulation, follow-up evaluation will be performed once every 6 months. Deep brain stimulation-related complications, such as dyskinesia, dysarthria, gait disorder, eye apraxia, depression, apathy and hypomania. Corresponding treatment methods will be administered. All these will be reported to the principal investigator and Institutional Review Board within 24 hours.

Data management According to the trial design, a table will be formulated for data collection. Collected data will be input into an electronic database by professional staff using a double-data entry strategy. Information accuracy will be checked when all recruited patients are followed up. The database will be locked by the researcher in charge and will not be altered. All information relating to this trial will be preserved by Department of Neurosurgery, Chinese PLA General Hospital of China. The electronic database will be fully disclosed to a professional statistician for statistical analysis.

Statistical analysis All data will be statistically analyzed by a statistician blinded to randomization using SPSS 18.0 software. The successive normally distributed variables will be expressed as the mean ± SD. The non-normally distributed variables will be expressed as median and quartile. Classification variables will be expressed as count and percentage. A paired t-test or Wilcoxon Matched-Pairs Signed-Rank Test will be used to compare the continuous variables of the primary and secondary outcome measures at each time point. The chi-square test or Fisher's exact test will be used to compare the classification variables. A P level of <0.05 will be accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnosis criteria of AD formulated by the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA);
* MMSE score 0-10 points;
* Age 40-80 years;
* Provision of signed informed consent.

Exclusion Criteria:

* Abnormal brain structure prior to surgery (tumor, cerebral infarction, intracranial hematoma)
* Complicated by other neurological system disorders, such as multiple sclerosis and epilepsy;
* Psychiatric disorders, such as anxiety, depression or drug-induced psychosis;
* Severe internal diseases, are taking respiratory system drugs, cardiovascular drugs, anticonvulsants or psychotropic drugs;
* Inability to tolerance clinical complications;
* Severe auditory and visual disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Six Patients with severe Alzheimer's disease (AD) scheduled to receive deep brain stimulation will be all recruited from the clinics and wards of Department of Neurosurgery, Chinese PLA General Hospital of China.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Deep brain stimulation-related disability rates | changes of baseline and month 1, month 6, month 12 after surgery
  To assess the effectiveness of deep brain stimulation in the treatment of Alzheimer's disease (AD).

SECONDARY OUTCOMES:
Clinical Dementia Rating(CDR) score | changes of baseline and month 1, month 6, month 12 after surgery
  The Clinical Dementia Rating(CDR) is 5-point scale used to characterize six domains (memory, orientation, judgment & problem solving, community affairs, home & hobbies and personal care) of the cognitive and functional performance of the aged (in particular AD patients). Patients are rated on dementia severity: 0 = normal, 0.5 = questionable dementia; 1 = mild dementia; 2 = moderate dementia; 3 = severe dementia.
The Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-Cog) | changes of baseline and month 1, month 6, month 12 after surgery
  The Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-Cog) scale is widely used for evaluating the severity of AD. ADAS-Cog consists of 12 components including word recall, naming, command, constructional praxis, ideational praxis, orientation, word recognition, remembering test instructions, spoken language ability, word finding difficulty, comprehension of oral language, and attention. The ADAS-Cog assesses multiple cognitive domains including memory, language, praxis, and orientation. ADAS-Cog score ranges from 0-75, with higher scores indicating more severe cognitive impairment.
Mini-Mental State Examination (MMSE) score | changes of baseline and month 1, month 6, month 12 after surgery
  Mini-Mental State Examination (MMSE) is one of the most influential cognitive screening tools worldwide. It consists of five dimensions including orientation (10 points), registration (3 points), attention and calculation (5 points), recall (3 points) and language and praxis (9 points). Educational attainment level-related dementia classification: illiterate: 5 points ≤ MMSE score ≤16 points; primary school: 8 points ≤ MMSE score ≤ 20 points; junior high school and above: 10 points ≤ MMSE score ≤ 24 points.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqi Mao, Ph.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu J, Liu B, Shang G, Feng Z, Yang H, Chen Y, Yu X, Mao Z. Efficacy and Safety of Bilateral Deep Brain Stimulation (DBS) for Severe Alzheimer's Disease: A Comparative Analysis of Fornix Versus Basal Ganglia of Meynert. CNS Neurosci Ther. 2025 Apr;31(4):e70285. doi: 10.1111/cns.70285. PMID 40243219
- [Derived] Mao ZQ, Wang X, Xu X, Cui ZQ, Pan LS, Ning XJ, Xu BX, Ma L, Ling ZP, Jia JJ, Yu XG. Partial improvement in performance of patients with severe Alzheimer's disease at an early stage of fornix deep brain stimulation. Neural Regen Res. 2018 Dec;13(12):2164-2172. doi: 10.4103/1673-5374.241468. PMID 30323149